CLINICAL TRIAL: NCT05152771
Title: Post Measles Subacute Sclerosing Panencephalitis (SSPE)and the Role of Ketogenic Diet, A Prospective Cohort Study
Brief Title: Role of Ketogenic Diet in SSPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: National Institute of Child Health, Karachi, Pakistan (Other Government)
Responsible Party: Principal Investigator, Dr Shahnaz Ibrahim, PROFESSOR, Aga Khan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-6491-19410.
Record Dates: First submitted 2021-11-03; First posted 2021-12-10 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: SSPE
Keywords: Ketogenic Diet; Progressive Neurological Disorder; Intractable Epilepsy
MeSH Terms: conditions — Subacute Sclerosing Panencephalitis; Drug Resistant Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet (Other): This will be a prospective cohort study. All families with children who have been newly diagnosed with confirmed SSPE (based on Dyken's Criteria) will be approached to start the low glycemic index diet (liberalized kind of KD). A thorough dietary history will be taken from the parents/caregivers, and they will be counseled by a trained dietitian on the diet, all pros and cons, and the format. After the verbal agreement, formal consent will be taken from the parent/ caregiver for initiation of the diet.
  Interventions: Other: KETOGENIC DIET

INTERVENTIONS:
Other: KETOGENIC DIET — This will be a prospective cohort study. All families with children who have been newly diagnosed with confirmed SSPE (based on Dyken's Criteria) will be approached to start the low glycemic index diet (liberalized kind of KD). A thorough dietary history will be taken from the parents/caregivers, and they will be counseled by a trained dietitian on the diet, all pros and cons, and the format. After the verbal agreement, formal consent will be taken from the parent/ caregiver for initiation of the diet.
  These patients are usually already admitted in the hospital for initial diagnosis and management. Therefore the initiation of the diet will be in the hospital during their admission if the parents/ caregivers agrees. A minimum of 2-3 days would be required to train the parents/caregivers.
  Other Names: LOW GLYCEMIC INDEX DIET

SUMMARY:
SSPE is a progressive neurodegenerative disorder occurring after measles infection and is potentially life-threatening.Measles infection remains endemic in Pakistan especially in the lower socioeconomic population where the vaccine coverage is low. The ketogenic diet has been used in a large number of diseases especially intractable epilepsies in children and also in certain neurodegenerative disorders like Parkinson's and Alzheimer's in adults. Some of the case reports from India and the USA have reported the beneficial results of ketogenic diet(KD) not only in the control of myoclonic jerks of SSPE but also in stopping and reversing the progress of the disease. There is a definite need to conduct a multi-center trial of KD to establish its effectiveness in SSPE.

At the Aga khan university, the investigators have an experienced team who have been using KD for the last 9 years for intractable epilepsy. At AKU the investigators currently have 4 patients on board for the past 4 months, with diagnosed SSPE on Low Glycemic Index Diet and showing some improvement in their seizure and motor control. Based on these reports, for a poor measles control country like Pakistan, there is a need to work further in order to establish evidence for KD therapy as a treatment for SSPE. The findings of the proposed study will serve as a hope for the improvement of quality of life of patients suffering from SSPE which is a devastating disease with almost 100% mortality .

DETAILED DESCRIPTION:
Methodology This will be a bi-center trial. The national institute of child health (NICH) will be a partner in this study along with Aga Khan University Hospital, Karachi. This study will be a nutritional research study looking at the role of the Ketogenic diet in improving seizures and overall disability in children with SSPE. LGIT will be the form of KD used for these patients.

All families with children who have been newly diagnosed with confirmed SSPE will be approached to start the low glycemic index diet,(liberalized kind of KD). They will be counseled on the disease and the diet regimen. all possible side effects and management will be discussed. The duration of follow-up will be for one year and there will be no potential cost incurred by the patient.

Patients will also be followed up by the physiotherapist at the physiotherapy department at AKU ( @ no cost)who will be supporting their motor rehabilitation. Investigations which include blood work and echo and ultrasound and EEGs will be done at regular intervals Sampling technique A consecutive sampling of all children who are diagnosed with SSPE will be used. A total of 26 children >2-<15 years will be enrolled over a period of two years.

ELIGIBILITY:
Inclusion Criteria:• All patients with a recent diagnosis of SSPE based on Dyken's criteria. Children aged ≥2 - ≤15 years.

• Having at least one member of the family residing with the patient who can read and understand directions in Urdu and /or Sindhi.

Exclusion Criteria:

* • Parents not agreeing to start the diet.

  * Age less than 2 years or over 15 years.
  * Patients who are already being given immune modulators.
  * Any other associated co-morbidity.
  * Patients having difficulty in swallowing and parents not allowing a nasogastric tube.
  * Totally uneducated family with no one who can read or write and understand directions in Urdu and/ or Sindhi.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Seizure control | for a period of 6 months .
  frequency and severity will be measured through a seizure record diary, daily number of seziures will be averaged over a month and monthly record will be evaluated as percentage increase or decrease in 3 months intervals

SECONDARY OUTCOMES:
cognitive Change , | base line, after 6 months of study then after and one year of study.
  checked by using Pedicat with 4 domains. Daily activities, Mobility and Social/Cognitive domains.The three functional skill domains are rated on a 4 point scale:
  1. Unable
  2. Hard
  3. A little hard
  4. Easy
  0.I don't know
  Responsibility:This domain has its own 5 point scale:
  1. Adult/caregiver has full responsibility;
  2. Adult/caregiver has most responsibility and child takes a little responsibility
  3. Adult/caregiver and child share responsibility about equally
  4. Child has most responsibility with a little direction, supervision or guidance from an adult/caregiver
  5. Child takes full responsibility without any direction, supervision or guidance from an adult/caregiver Two types of score will calculate: normative scores and scaled scores. The normative score is based on the child's chronological age. Scaled score provides a way to look at current functional skills and progress in skills over times (compare the child towards itself).
behavioral Change | base line, after 6 months of study then after and one year of study
  this will be checked by using modified Ashworth scales.MODIFIED ASHWORTH The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform.
  scoring 0 No increase in tone 1 slight increase in tone giving a catch when slight increase in muscle tone, manifested by the limb was moved in flexion or extension.
  1+ slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM ) 2 more marked increase in tone but more marked increased in muscle tone through most limb easily flexed 3 considerable increase in tone, passive movement difficult 4 limb rigid in flexion or extension
motor developmental Change | base line, after 6 months of study then after and one year of study
  this will be checked by , Modified Rankin and GMFM Modified Rankin Scale Score Description 0 No symptoms at all
  1. No significant disability despite symptoms
  2. Slight disability
  3. Moderate disability
  4. Moderately severe disability
  5. Severe disability
  6. Dead GMFM There is a scoring system with each item scored as 0, 1, 2, 3, or "not tested". A scoring key of 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed, is used; however parameters such as distance, time, support provided, accuracy, counts, and tasks will determine specific item scores. Items that a child refuses to attempt despite reason they may be able to perform at least partially or items not administered are scored as 'not tested'.
  The scoring system of the GMFM is a four-point scale that consists of 66 items divided into five dimensions of gross motor function:(a) lying and rolling, (b) sitting, (c) crawling and kneeling, (d) standing, and (e) walking, running and jumping.

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz H Ibrahim, MBBS ;FCPS, Principal Investigator — AKU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rafique A, Amjad N, Chand P, Zaidi SS, Rana MS, Ahmed K, Ibrahim S. Subacute sclerosing panencephalitis: clinical and demographic characteristics. J Coll Physicians Surg Pak. 2014 Aug;24(8):557-60. PMID 25149833
- [Result] Ibrahim SH, Amjad N, Saleem AF, Chand P, Rafique A, Humayun KN. The upsurge of SSPE--a reflection of national measles immunization status in Pakistan. J Trop Pediatr. 2014 Dec;60(6):449-53. doi: 10.1093/tropej/fmu050. Epub 2014 Sep 16. PMID 25232151
- See also: Jafri SK, Kumar R, Ibrahim SH. Subacute sclerosing panencephalitis - current perspectives. Pediatric Health Med Ther. 2018;9:67-71 — http://doi.org/10.2147/PHMT.S126293